CLINICAL TRIAL: NCT00583323
Title: Diphenoxylate / Atropine to Decrease Bowel Activity During F-18 FDG PET
Brief Title: Diphenoxylate / Atropine to Decrease FDG Activity During F-18 FDG PET
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Val J. Lowe, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Diagnostic
Other Study IDs: 2051-02
Record Dates: First submitted 2007-12-20; First posted 2007-12-31 (Estimated); Last update posted 2014-08-21 (Estimated); Status verified 2014-08

CONDITIONS: Lymphoma
MeSH Terms: conditions — Lymphoma | interventions — atropine sulfate-diphenoxylate hydrochloride drug combination; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Lomotil given
  Interventions: Drug: Lomotil
- 2 (Placebo Comparator): Normal Saline given
  Interventions: Other: Normal saline

INTERVENTIONS:
Drug: Lomotil — Orally 10ml of Lomotil
  Arms: 1
Other: Normal saline — 10 ml orally
  Arms: 2

SUMMARY:
2-[18F]-fluoro-2-deoxyD-glucose positron emission tomography (FDG PET) has proven to be a valuable clinical tool for the staging and surveillance of lymphoma.1-6 Occasionally, lymph nodes in the mesentery and retroperitoneum can be difficult to distinguish from normal bowel activity on PET scans despite three-plane and cine maximal image projection (MIP) imaging. This uncertainty limits the clinical usefulness of PET in some cases of lymphoma.7-8 In addition, bowel activity can also hinder interpretation of PET scans in other types of solid tumors including melanoma and colorectal cancer.6,9,10 Our goal is to determine how well diphenoxylate/atropine 5mg/0.05mg (Lomotil) decreases bowel activity and how this decrease impacts clinical decision-making, specifically for lymphoma staging and surveillance. This is a prospective, randomized, double-blinded study involving 60 patients undergoing PET scans for newly diagnosed or recurrent, untreated lymphoma.

ELIGIBILITY:
Inclusion Criteria

* Males and females 18 years of age or older
* Subjects pre-scheduled for clinically-indicated PET scan
* Subjects with newly diagnosed or recurrent untreated disease (lymphoma) based on abdominal and/or pelvic adenopathy or masses on CT within 6 months of PET scan Exclusion Criteria
* Allergy to Lomotil (Diphenoxylate hydrochloride, Atropine sulfate)
* Subjects with one or more episodes of diarrhea within 24 hours prior to PET scan
* Women who are breast-feeding
* Subjects with a history of severe liver disease, jaundice, dehydration, or narrow-angle glaucoma

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2003-02; Primary Completion 2005-09 (Actual); Study Completion 2005-09 (Actual)

PRIMARY OUTCOMES:
Reduction of bowel activity | 1hour

SECONDARY OUTCOMES:
Reduction of stomach activity | 1 hour